CLINICAL TRIAL: NCT03953937
Title: Classification and Comparison of Early-onset and Late-onset Idiopathic Chronic Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Department, Changhai Hospital
Other Study IDs: ICP-1
Record Dates: First submitted 2019-05-08; First posted 2019-05-17 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pancreatitis; Idiopathic Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICP cohort: Patients with idiopathic pancreatitis

SUMMARY:
Classification of early-onset idiopathic chronic pancreatitis (EOICP) and late-onset idiopathic chronic pancreatitis (LOICP) was proposed based on bimodal distribution of age at onset of idiopathic chronic pancreatitis (ICP). However, studies of larger populations prove it may be normal distribution. Therefore, the aim of the study is to find what the distribution of age at onset of ICP is and whether the classification of EOICP and LOICP is meaningful.

DETAILED DESCRIPTION:
Idiopathic chronic pancreatitis (ICP) patients admitted to the investigator's center from January 2000 to December 2013 were enrolled. Characteristics were compared between early-onset idiopathic chronic pancreatitis (EOICP) and late-onset idiopathic chronic pancreatitis (LOICP) patients. Cumulative rates of diabetes mellitus, steatorrhea, pancreatic stone, pancreatic pseudocyst (PPC), biliary stricture, and pancreatic cancer after the onset and the diagnosis of ICP were calculated, respectively. Different cut-off values for age at onset of ICP were set to classify EOICP and LOICP. Then differences of clinical courses between EOICP and LOICP were compared when classified by distinct cut-off values.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic chronic pancreatitis according to Asia-Pacific consensus

Exclusion Criteria:

* Pancreatic cancer diagnosed within 2 years after the diagnosis of chronic pancreatitis
* Groove pancreatitis
* Autoimmune pancreatitis
* Chronic pancreatic patients with identified etiologies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Idiopathic chronic pancreatitis patients in China
Sampling Method: Probability Sample
Enrollment: 1633 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of age at onset of idiopathic chronic pancreatitis | December 31, 2013
  Identify the distribution of age at onset of idiopathic chronic pancreatitis.
Basic characteristics of early-onset idiopathic chronic pancreatitis and late-onset idiopathic chronic pancreatitis | December 31, 2013
  Identify respective ratio of patients with male gender and patients with smoking history in early-onset idiopathic chronic pancreatitis and late-onset idiopathic chronic pancreatitis in traditional classification (traditional classification: age at onset of idiopathic chronic pancreatitis<35 years old as early-onset idiopathic chronic pancreatitis; age at onset of idiopathic chronic pancreatitis>35 years old as late-onset idiopathic chronic pancreatitis).

SECONDARY OUTCOMES:
Basic characteristics of early-onset idiopathic chronic pancreatitis and late-onset idiopathic chronic pancreatitis with different cut-off values for age at onset of idiopathic chronic pancreatitis | August 31, 2019
  Identify respective ratio of patients with male gender and patients with smoking history in early-onset idiopathic chronic pancreatitis and late-onset idiopathic chronic pancreatitis with different cut-off values for age at onset of idiopathic chronic pancreatitis.
Diabetes mellitus | August 31, 2019
  Evaluate incidence and cumulative incidence of endocrine insufficiency developed in early-onset and late-onset idiopathic chronic pancreatitis patients with different cut-off values for age at onset of idiopathic chronic pancreatitis.
Steatorrhea | August 31, 2019
  Evaluate incidence and cumulative incidence of exocrine insufficiency developed in early-onset and late-onset idiopathic chronic pancreatitis patients with different cut-off values for age at onset of idiopathic chronic pancreatitis.
Pancreatic pseudocyst | August 31, 2019
  Evaluate incidence and cumulative incidence of pancreatic pseudocyst developed in early-onset and late-onset idiopathic chronic pancreatitis patients with different cut-off values for age at onset of idiopathic chronic pancreatitis.
Common bile duct stricture | August 31, 2019
  Evaluate incidence and cumulative incidence of common bile duct stricture developed in early-onset and late-onset idiopathic chronic pancreatitis patients with different cut-off values for age at onset of idiopathic chronic pancreatitis.
Pancreatic cancer | August 31, 2019
  Evaluate incidence and cumulative incidence of pancreatic cancer developed in early-onset and late-onset idiopathic chronic pancreatitis patients with different cut-off values for age at onset of idiopathic chronic pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Doctor, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China